CLINICAL TRIAL: NCT04809181
Title: Azacitidine in Combination With Venetoclax Treatment for Prevention of Relapse in MRD Positive Post Allogeneic Hematopoietic Stem Cell Transplantation Acute Myelogenous Leukemia/ Myelodysplastic Syndrome Patients
Brief Title: Azacitidine in Combination With Venetoclax Treatment for MRD Positive Post Allo-HSCT AML/MDS Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Sir Run Run Shaw Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); Yinzhou Hospital Affiliated to Medical School of Ningbo University (Other); Jinhua Central Hospital (Other); Taizhou Hospital (Other); Union hospital of Fujian Medical University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yi Luo, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU-HSCT-AZA02
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hematologic Malignancy; Stem Cell Transplant Complications
Keywords: Allogeneic Hematopoietic stem cell transplantation; Micro residual disease; Azacitidine; Venetoclax; Relapse
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD positive AML/MDS patients after allogeneic hematopoietic stem cell transplantation (Experimental): MRD positive AML/MDS patients after allogeneic hematopoietic stem cell transplantation
  Interventions: Drug: Azacitidine in Combination With Venetoclax

INTERVENTIONS:
Drug: Azacitidine in Combination With Venetoclax — Azacitidine in combination with venetoclax

SUMMARY:
In patients with MRD-positive patients after AML/MDS allogeneic hematopoietic stem cell transplantation, azacytidine combined with venetoclax may be effective in eliminating micro residual diseases, reducing the risk of relapse, and ultimately improving long-term survival.The primary purpose of this study was to explore an effective protocol to reduce the risk of relapse in patients with MRD positive after allogeneic hematopoietic stem cell transplantation for AML/MDS.

DETAILED DESCRIPTION:
The technology of Allogeneic Hematopoietic stem cell transplantation (allo-HSCT) has been continuously improved, relpase is still the leading cause of death after allo-HSCT. Monitoring of micro residual disease (MRD) after allogeneic HSCT provides a risk stratification of relpase risk in patients after transplantation.There is an urgent need to find an effective intervention plan for patients with MRD positive after transplantation, in order to reduce the risk of relapse after transplantation and improve long-term survival.The combination of demethylated drugs with venetoclax has shown promising results in clinical trials in AML patients who cannot tolerate induction chemotherapy.In patients with MRD-positive patients after AML/MDS allo-HSCT, azacytidine combined with venetoclax may be effective in eliminating small residual diseases, reducing the risk of relapse, and ultimately improving long-term survival.The primary purpose of this study was to explore an effective protocol to reduce the risk of relapse in patients with MRD positive after allo-HSCT for AML/MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 years old and 65 years old.
2. Patients with AML or MDS diagnosed according to WHO diagnostic criteria.
3. Patients who received allogeneic hematopoietic stem cell transplantation and achieved complete remission.
4. MRD was positive after transplantation, MFC > 0.1% and / or fusion gene and gene mutation (WT1 > 0.6%, AML1-ETO > 0.4%, others >1%).
5. ECOG body status score 0-2.
6. Patients with expected survival time >=3 months.
7. Good organ function level: ANC (neutrophil absolute value >=1.0x10^9/L; PLT >=30x10^9/L; HB >=80g/L; Tibil <=1.5 ULN; ALT / AST <=2.5 ULN; bun / Cr <=1.5 ULN; LVEF >=50%).
8. Patients who have received any anti-tumor treatment (including radiotherapy, chemotherapy, surgery or molecular targeted treatment) for more than 4 weeks from the end of the previous treatment.
9. Patients with no GVHD and no previous history of 3 or more degrees of aGVHD. 10. Patients who voluntarily participate in the clinical trial, understand the research procedure and can sign the informed consent in writing.

Exclusion Criteria:

1. Patients with severe cardiac insufficiency and EF lower than 60%; or patients with severe arrhythmia who could not tolerate super pretreatment.
2. Patients with activity of aGVHD or extensive cGVHD.
3. Patients with BCR/ABL positive.
4. Patients who were previously known to be resistant to azacytidine or dessicabine or venetoclax.
5. In patients with severe pulmonary insufficiency (obstructive and / or restrictive ventilation disorders), the researchers evaluated the patients who could not tolerate the super pretreatment scheme.
6. Patients with severe liver function impairment and liver function indexes (alt, TBIL) more than 3 ULN were evaluated as intolerant of super pretreatment.
7. In patients with severe renal insufficiency, the renal function index (CR) is more than 2 times of the upper limit of the normal value (ULN), or the 24-hour creatinine clearance rate (CR) is less than 50ml / min, the researchers evaluated that they could not tolerate the super pretreatment scheme.
8. In patients with severe active infection, the researchers evaluated that they could not tolerate the pretreatment.
9. Patients who had allergic reactions or serious adverse reactions in the previous use of pretreatment related drugs could not be included in the study.
10. Patients with hematological recurrence (bone marrow smear: proportion of primordial cells >=5%) or any extramedullary recurrence.
11. Other reasons why the researchers could not be selected.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival | 2 year
  relapse-free survival

SECONDARY OUTCOMES:
overall survival | 2 year
  overall survival
graft-versus-host disease -free relapse-free survival | 2 year
  graft-versus-host disease -free relapse-free survival
cumulative incidence of aGVHD | 100 days
  cumulative incidence of aGVHD
cumulative incidence of cGVHD | 2 year
  cumulative incidence of cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (1):
- The first Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No